CLINICAL TRIAL: NCT00981006
Title: Hybrid Biotherapy Involving Autologous Human Cardiac Stem Cell Transplantation Combined With the Controlled Release of bFGF Using a Gelatin Hydrogel Sheet to Treat Severe Refractory Heart Failure With Chronic Ischemic Cardiomyopathy
Brief Title: AutoLogous Human CArdiac-Derived Stem Cell to Treat Ischemic cArdiomyopathy (ALCADIA)
Acronym: ALCADIA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Naofumi Takehara (Other)
Collaborators: National Cerebral and Cardiovascular Center, Japan (Other); Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other); Asahikawa Medical College (Other)
Responsible Party: Sponsor-Investigator, Naofumi Takehara, Assistant Professor, Kyoto Prefectural University of Medicine
Organization: Kyoto Prefectural University of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRICAD0910; TRICAD0806 (Registry Identifier: TRI); NCT01697033 (obsolete NCT alias)
Record Dates: First submitted 2009-09-19; First posted 2009-09-21 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Congestive Heart Failure; Ischemic Cardiomyopathy; Ventricular Dysfunction
Keywords: ischemic cardiomyopathy (ICM)
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction | interventions — KCB-1 protein, recombinant; Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- human cardiac stem cell therapy (Experimental): single administration of 0.5 million cells/kg(patient body weight) of human cardiac stem cells and 200 microgram of bFGF at coronary artery bypass grafting (CABG)
  Interventions: Procedure: human cardiac stem cells

INTERVENTIONS:
Procedure: human cardiac stem cells — Single intramyocardial Injection of autologous hCSCs : 20 cites of infarcted myocardium Implantation of gelatin hydrogel sheet incorporating bFGF: 200 microgram. CABG surgery.
  Other Names: human cardiac stem cell (hCSC); human recombinant basic fibroblast growth factor (bFGF); coronary artery bypass grafting (CABG)

SUMMARY:
The aim of this study is to evaluate the safety and efficacy on the transplantation of autologous human cardiac-derived stem cells (hCSCs) with the controlled release of basic fibroblast growth factor (bFGF) to severe refractory heart failure patients with chronic ischemic cardiomyopathy concordance with reduced left ventricular dysfunction (15%≦LVEF≦35%).

DETAILED DESCRIPTION:
Autologous human stem or progenitor cells of different lineage have been subjected to clinical trials in the past to treat patients with ischemic cardiomyopathy. Although human stem or progenitor cells transplantation had functional benefits in the recovery in experimental myocardial infarction, the major barrier limiting its clinical application is the death of the most of the transplanted cells and poor cardiac differentiation in the host environment. Using the identical technique as clonally cell isolation from experimental animals, we generated human cardiac-derived stem cell (hCSC) enriched Es-marker genes with mesenchymal features. hCSCs included in cell populations accelerating proliferation in the presence of basic fibroblast growth factor (bFGF) on plastic plates are generated from human heart tissues through endomyocardial biopsy. Giving a patient their own hCSCs is an investigational procedure that has been approved by the committee of the Ministry of Health, Labour, and Welfare of Japan for this study. hCSCs have excellent potential to proliferate and regenerate to cardiomyocyte compared with other cells, e.g. myoblasts, bone marrow mononuclear cells and bone marrow stem cells, already evaluated in preliminary experiments on the repair of injured heart muscle. bFGF possesses properties to promote stem cell proliferation, and formation of sufficient microvascular network created by bFGF is critical for long-term survival of transplanted donor cells. This will be the first trial on the use of autologous hCSCs for the treatment of refractory heart failure with chronic ischemic cardiomyopathy. This trial is translational pilot study for looking into the safety and efficacy on the use of autologous hCSCs with the controlled release of bFGF using a gelatin hydrogel sheet.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of ischemic cardiomyopathy

   * Ischemic cardiomyopathy with old myocardial infarction due to coronary artery atherosclerotic disease.
2. Age: 20 to 80 years old
3. left ventricle (LV) dysfunction : An ejection fraction (EF)≧15%, and ≦35% assessed by echocardiography
4. Refractory heart failure: American Heart Association (AHA)/American College of Cardiology (ACC)heart failure Stage D
5. Heart failure symptom: New York Heart Association (NYHA) Class III or IV
6. An indication for CABG:A myocardial ischemia according to major coronary artery stenosis (>75%)
7. Viability in the infarct area as measured by cardiac delayed hyperenhancement magnetic resonance imaging (MRI)

   * Infarct area affecting >2 contiguous LV segments in a 18-segment model
   * The number of segments which transmural extent of hyperenhancement more than 51% is less than one.

     * Ex1. infarct area with or without bypass graft.
     * Ex2. no correlation with graft number.
     * Ex3. in case of multiple myocardial infarction, an indication for larger in infarct volume.
8. written informed consent

Exclusion Criteria:

1. New onset of myocardial infarction or unstable angina within 28 days prior to study entry
2. Indication for surgical ventricular reconstruction or mitral valve repair *1
3. Contraindication for endomyocardial biopsy *2
4. Evidence for malignant disease within 3 years prior to study entry
5. Chronic hemodialysis
6. Liver Cirrhosis (ICGR 15 >30%)
7. Uncontrollable diabetes mellitus (HbA1c>8.0)
8. Maximum diameter of Aortic aneurysm more than 5.5 cm.(including dissecting aneurysm)
9. Cardiogenic shock
10. Active infection (including cytomegalovirus infection)
11. Drug or alcoholic dependency
12. Positive for HIV antigen
13. Active bleeding state (gastric ulcer, cerebral bleeding, etc.)
14. Gelatin allergy *3
15. Chromosomal abnormality

    * 1 an indication for LV aneurysmectomy; patients with over 2 segments of dyskinesis area
    * 2 contra-indication for endomyocardial biopsy

      * cardiogenic shock
      * end-stage or uncontrollable congestive heart failure without continues infusion of catecholamine
      * complete or mobitz type atria-ventricular block
    * 3 The screening of gelatin allergy is necessary for all patients by gelatin patch test and gelatin-immunoglobulin E.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the safety of autologous cardiac-derived stem cells administered by intra-myocardial injection with the controlled release of bFGF in severe refractory heart failure patients with chronic ischemic cardiomyopathy. | 12 month

SECONDARY OUTCOMES:
The secondary objective is to demonstrate the safety of autologous cardiac-derived stem cells administered by intra-myocardial injection with the controlled release of bFGF in severe refractory heart failure patients with chronic ischemic cardiomyopathy. | 12month

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Matsubara, MD,PhD, Principal Investigator — Kyoto Prefectural University School of Medicine
Locations (2):
- Japan (2):
  - Kyoto Prefectural University School of Medicine, Kyoto, Kajii-cho 465, Hirokoji-agaru, Kawaramachi-dori,kamikyoku
  - National Cardiovascular Center, Osaka

REFERENCES:
- [Background] Takehara N, Tsutsumi Y, Tateishi K, Ogata T, Tanaka H, Ueyama T, Takahashi T, Takamatsu T, Fukushima M, Komeda M, Yamagishi M, Yaku H, Tabata Y, Matsubara H, Oh H. Controlled delivery of basic fibroblast growth factor promotes human cardiosphere-derived cell engraftment to enhance cardiac repair for chronic myocardial infarction. J Am Coll Cardiol. 2008 Dec 2;52(23):1858-1865. doi: 10.1016/j.jacc.2008.06.052. PMID 19038683
- [Background] Tateishi K, Ashihara E, Takehara N, Nomura T, Honsho S, Nakagami T, Morikawa S, Takahashi T, Ueyama T, Matsubara H, Oh H. Clonally amplified cardiac stem cells are regulated by Sca-1 signaling for efficient cardiovascular regeneration. J Cell Sci. 2007 May 15;120(Pt 10):1791-800. doi: 10.1242/jcs.006122. PMID 17502484
- [Background] Tateishi K, Ashihara E, Honsho S, Takehara N, Nomura T, Takahashi T, Ueyama T, Yamagishi M, Yaku H, Matsubara H, Oh H. Human cardiac stem cells exhibit mesenchymal features and are maintained through Akt/GSK-3beta signaling. Biochem Biophys Res Commun. 2007 Jan 19;352(3):635-41. doi: 10.1016/j.bbrc.2006.11.096. Epub 2006 Nov 27. PMID 17150190
- [Derived] Chimenti I, Gaetani R, Forte E, Angelini F, De Falco E, Zoccai GB, Messina E, Frati G, Giacomello A. Serum and supplement optimization for EU GMP-compliance in cardiospheres cell culture. J Cell Mol Med. 2014 Apr;18(4):624-34. doi: 10.1111/jcmm.12210. Epub 2014 Jan 20. PMID 24444305
- See also: Click here for more information about this study — http://www.f.kpu-m.ac.jp/k/med2/index.html